CLINICAL TRIAL: NCT05911659
Title: Ndividualized and Combined Effects of Diabetes and Smoking on the Antiplatelet Activity of Ticagrelor in Acute Myocardial Infarction Patients Undergoing Primary PCI
Brief Title: Individualized and Combined Effects of Diabetes and Smoking on the Antiplatelet Activity of Ticagrelor in Acute Myocardial Infarction Patients Undergoing Primary PCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mina Wageh Mohareb (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor-Investigator, Mina Wageh Mohareb, Professor, Cairo University
Organization: Cairo University (Other)
Other Study IDs: Al-Azhar University
Record Dates: First submitted 2023-06-10; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Individualized and Combined Effects of Smoking and Diabetes on the Antiplatelet Activity in Patients Undergoing Primary Percutaneous Coronary Intervention
MeSH Terms: interventions — Ticagrelor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Non smokers- non diabetic patients
  Interventions: Drug: Ticagrelor
- smokers non diabetic patients
  Interventions: Drug: Ticagrelor
- non smokers diabetic patients
  Interventions: Drug: Ticagrelor
- smokers diabetic patients
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — Patients with acute coronary syndromes undergo primary PCI and administered 180 mg loading dose ticagrelor before PCI
  Other Names: Primary percutaneous coronary intervention (PCI)

SUMMARY:
Background:Diabetes and smoking are common factors found to increase platelet reactivity in patients undergoing primary PCI. Objective: Compare the individualized and combined effects of smoking and diabetes on the antiplatelet activity in patients undergoing primary PCI. Methods: sixty patients were recruited in this study. Patients were allocated to one of four groups according to the diabetes and smoking status. Non smokers- non diabetic patients, smokers non diabetic patients, non smokers diabetic patients, and smokers diabetic patients, 15 patients in each group. All patients received 180 mg ticagrelor before PCI. Platelet reactivity index(PRI) and maximum platelet aggregation were measured 24 hours after ticagrelor loading dose for each patient as indicators for antiplatelet efficacy. PRI and/or MPA values > 50% were defined as high platelet reactivity.

ELIGIBILITY:
Inclusion Criteria:

Acute coronary syndrome (ACS) undergoing PCI

Exclusion Criteria:

Patients who had a history of severe bleeding, serious bleeding tendency, history of intracranial hemorrhage, signs of active bleeding, thrombocytopenia, uncontrolled hypertension, hypersensitivity to the used drugs (clopidogrel or ticagrelor), concomitant use of strong CYP inducers or inhibitors, and/or severe liver disorders were excluded from the study.

Patients with previous history of coronary artery disease, previous PCI or patients administering other antiplatelets were excluded from the current study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with ACS undergoing PCI
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Platelet Reactivity Index and maximum platelet aggregation | 24 hours after PCI
  Platelet aggregation indicator

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine of girls, Cardiology department, Al-Azhar University in Cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No